CLINICAL TRIAL: NCT06911216
Title: A Multiple-Dose Pharmacokinetics (PK) Study of STN1013800 in Healthy Adults
Brief Title: A Pharmacokinetics (PK) Study in Healthy Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101380004CN
Record Dates: First submitted 2025-03-11; First posted 2025-04-04 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Blepharoptosis
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STN1013800 ophthalmic solution (Experimental): 0.1% STN1013800 ophthalmic solution administered once daily (QD) for 7 days
  Interventions: Drug: STN1013800 ophthalmic solution

INTERVENTIONS:
Drug: STN1013800 ophthalmic solution — Investigational Product: 0.1% STN1013800 ophthalmic solution once daily (QD) (9AM ± 60 min), one drop for each eye

SUMMARY:
This is to characterize STN1013800 active ingredient bioavailability following multiple-dose ocular administration of STN1013800 to both eyes in healthy adults.

It is a PK study with screening period of up to 28 days + dosing period of 7 days + Follow-up period of 2 days.

At present, there are no medicines for the treatment of acquired blepharoptosis in China.

Therefore, efficacy and safety phase III study is also currently being conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to understand and sign the informed consent form approved by the independent ethics committee.
2. Age: 18～45 years old; male and female genders.
3. Best corrected visual acuity≥1.0 with no diagnosed ocular or rheumatologic disorders (e.g. dry eyes) that may affect vision.
4. Current non-smokers who have not used tobacco or nicotine in any form (including non-nicotine vaping/electronic cigarette products) at least 6 months prior to Day -1.
5. Weigh at least 50 kg and have a standard Body Mass Index (BMI) (19-24, Boundary containing value) at the time of screening.
6. Female volunteers, for pregnancy avoidance/prevention, the subject should be sterile, postmenopausal or approved methods of contraception.
7. Male volunteers for pregnancy avoidance/prevention of subject's female partner (if any), the subject should be sterile, not sexually active, or using approved methods of contraception.
8. Judged by the Investigator to be healthy based on the medical history and screening procedures (physical examination, 12-lead ECG, vital signs, and laboratory test results)
9. Negative test for selected drugs of abuse, cotinine and alcohol at the Screening visit and on Day -1.
10. Negative serum hepatitis panel, negative Human Immunodeficiency Virus (HIV), and treponema pallidum antibody tests at the Screening visit.
11. Negative pregnancy test for females of childbearing potential at the Screening visit and on Day -1.
12. Understands the study requirements and willing to participate in the study.

Exclusion Criteria:

1. Participation in any other investigational study drug trial in which receipt of an investigational study drug or device occurred within 30 days prior to Day -1.
2. Contact lenses wearing during dose administration.
3. Use of any over-the-counter (OTC), non-prescription preparations (including multivitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) within the 14 days or 5 half-lives, whichever is longer, prior to Day -1.
4. Use of any prescription medications within the 14 days or 5 half-lives, whichever is longer prior to Day -1.
5. History or presence of any significant metabolic, allergic, cardiovascular, pulmonary, hepatic, renal, hematologic (including bleeding disorders), gastrointestinal (including peptic ulcer disease, gastritis or bleeding diathesis, excluding appendectomy or hernia repair), endocrine, immunologic, dermatologic, muscular, genitourinary, neurological, ophthalmologic, psychiatric, neoplastic, or other disease, that, in the opinion of the investigator, could interfere with the course of the study or expose the subject to undue risk by participating in this study.
6. Known hypersensitivity or idiosyncratic reaction to oxymetazoline or any related products (including excipients of the formulation) as well as severe hypersensitivity to any drugs.
7. History of cancer within the past 5 years, except for basal cell carcinoma with documentation of a 6-month remission at the Screening visit.
8. Any clinically significant illness in the previous 28 days before Day-1.
9. Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort), in the previous 28 days before Day-1.
10. Current use of a beta blocker or tricyclic antidepressant.
11. Any history of ocular hypertension or glaucoma; heart disease, angina, arteriosclerotic disease, or irregular heartbeat; hyperthyroidism; diabetes mellitus; poor peripheral venous access.
12. Any history of tuberculosis and/or prophylaxis for tuberculosis.
13. Urinary hesitancy or retention from prostatic hypertrophy.
14. Receipt or donation of any blood products within 3 months prior to Day-1.
15. History or presence of alcoholism or drug abuse or dependence (addiction), as determined at the discretion of the Investigator, within the past 2 years.
16. Seated (after at least 5 minutes in a sitting position) systolic blood pressure >140 mmHg or <90 mmHg or a diastolic blood pressure >90 mmHg at the Screening visit (blood pressure may be re-tested up to twice in the seated position at intervals of at least 5 minutes; the pressure elevation is considered sustained if either the systolic or diastolic pressure exceeds the states limits after 3 assessments).
17. Pulse rate at rest (after at least 5 minutes in a sitting position) of <60 bpm or >100 bpm at the Screening visit.
18. History of clinically significant abnormal ECG findings or a Screening ECG including but not limited to a second- or third-degree AV; QRS >120 milliseconds (msec); QTcF >450 msec for males or QTcF >470 msec for females; PR interval >240 msec; or any rhythm other than normal sinus rhythm that is deemed clinically significant by the Investigator.
19. Hospitalization during the 3 months prior to the Screening visit except for minor scheduled outpatient procedures.
20. In the Investigator's opinion, have been on an abnormal diet (for whatever reason) during the 28 days prior to Day-1.
21. For male subjects: intent to donate sperm from the first drug administration until 30 days after the last dose administration.
22. Any acute or chronic medical or psychiatric condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study.
23. Periocular neurotoxin (e.g., Botox, Xeomin, Dysport, Myobloc) injections within 3 months prior to Day -1 and during the study.
24. Taken any monoamine oxidase inhibitor (MAOIs) (e.g., isocarboxazid, phenelzine, tranylcypromine) within 14 days prior to Day-1 and during the study.
25. Topical application of bimatoprost (i.e., Latisse®) to the eyelashes within 7 days prior to Day-1 and during the study.
26. Topical ophthalmic medications (including but not limited to anti-allergy [e.g., antihistamines], dry eye [i.e.,Restasis®, Xiidra®], antimicrobial drugs [e.g., antibiotics and antivirals], and anti-inflammatory drugs [including nonsteroidal anti-inflammatory drugs (NSAIDs) and steroids] other than the assigned study medication within 7 days prior Day-1 and during the study. All topical antiglaucoma medications are prohibited.
27. Intravitreal injections (e.g., Lucentis®, Eylea®, Avastin®, Triesence®) within 7 days prior to Screening visit and during the study.
28. Current punctal plugs or placement of punctal plugs during the study.
29. Use of any OTC vasoconstrictor/decongestant eye medication (e.g., Visine® L.R.®) or any ophthalmic or non-ophthalmic α-adrenergic agonist including OTC products (e.g., Afrin®) within 7 days prior Day-1 and during the study. Artificial tears are allowed up to 24 hours prior to first drug administration.
30. Any consistent or intermittent use of oxymetazoline containing medications, including oxymetazoline nasal spray or oral products within 30 days prior to Screening visit and during study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
PK (Pharmacokinetic) parameter to measure: Cmax | Day 1, 5, 6, and 7
  Blood samples will be collected on Day 1, Day 5, Day 6, and Day 7. Cmax - Peak concentration
PK parameter to measure: Cmin | Day 1, 5, 6, and 7
  Blood samples will be collected on Day 1, Day 5, Day 6, and Day 7. Cmin - Minimum concentration
PK parameter to measure: Tmax | Day 1, 5, 6, and 7
  Blood samples will be collected on Day 1, Day 5, Day 6, and Day 7. Tmax - Peak time
PK parameter to measure: AUC0-24h | Day 1, 5, 6, and 7
  Blood samples will be collected on Day 1, Day 5, Day 6, and Day 7. AUC0-24h - The area under the drug-time curve for the quantifiable time period from 0 to 24 hours after drug administration.
PK parameter to measure: AUC0-36h | Day 1, 5, 6, and 7
  Blood samples will be collected on Day 1, Day 5, Day 6, and Day 7. AUC0-36h - The area under the drug-time curve from 0 to 36 hours after drug administration
PK parameter to measure: AUCinf | Day 1, 5, 6, and 7
  Blood samples will be collected on Day 1, Day 5, Day 6, and Day 7. AUCinf - The area under the drug-time curve from 0 to infinity after drug administration
PK parameter to measure: kel | Day 1, 5, 6, and 7
  Blood samples will be collected on Day 1, Day 5, Day 6, and Day 7. kel - Elimination rate constant. The negative of the slope value obtained by taking the logarithm of the plasma concentration in the vanishing phase of the time curve and performing linear regression on time obtained.
PK parameter to measure: t½ | Day 1, 5, 6, and 7
  Blood samples will be collected on Day 1, Day 5, Day 6, and Day 7. t½ - Elimination half-life

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital, Capital Medical University, Beijing, China